CLINICAL TRIAL: NCT03628534
Title: Saline Enhanced Radiofrequency (SERF) VT Ablation Early Feasibility Study (EFS)
Brief Title: SERF VT Ablation Early Feasibility Study (EFS)
Acronym: SERF VT EFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thermedical, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-100; 1R44HL132746-01A1 (NIH)
Record Dates: First submitted 2018-07-26; First posted 2018-08-14 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Ventricular Tachycardia; Arrythmia; Heart Diseases; Cardiovascular Diseases
Keywords: Cardiac Arrhythmia; Ventricular Tachycardia; Arrhythmia; Pathological processes
MeSH Terms: conditions — Tachycardia, Ventricular; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes

STUDY DESIGN:
Intervention Model Description: Thermedical SERF Ablation System and Durablate Catheter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- single arm (Experimental): Ablation of ventricular tachycardia with a saline-enhanced radiofrequency ablation catheter
  Interventions: Device: Saline Enhanced Radiofrequency (SERF) ablation

INTERVENTIONS:
Device: Saline Enhanced Radiofrequency (SERF) ablation — Ablation of ventricular tachycardia with a saline-enhanced radiofrequency ablation catheter
  Other Names: Durablate Catheter and Thermedical Ablation System

SUMMARY:
This is an early feasibility, non-randomized, open-label, single group, interventional study to be conducted in up to 20 US subjects to evaluate the technical feasibility of the Durablate Catheter and Thermedical Ablation System to eliminate or control sustained, monomorphic ventricular tachycardia (VT) in patients with VT refractory to drug and conventional catheter ablation with acceptable procedural safety.

DETAILED DESCRIPTION:
The purpose of this study is to gather information on the technical feasiability and safety of a needle ablation catheter called the Durablate™ Saline Enhanced Radiofrequency (SERF) catheter. This catheter is being studied to treat ventricular tachycardia (VT) in patients who have already been treated with medicine, have an Implantable Cardioverter Defibrillator (ICD) and had an ablation procedure to treat their VT but continue to experience VT despite these treatments. A VT ablation procedure is done by finding the abnormal heart tissue that's causing the VT and applying energy with the tip of an ablation catheter to the area to create a scar or destroy the tissue that causes the VT. The SERF catheter being used in this study uses a needle to deliver heated saline (salt water) and radiofrequency energy deeper into the heart tissue that is causing the VT than a standard ablation catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has sustained, monomorphic VT
2. Subject has recurrent, symptomatic VT
3. Subject has drug refractory or drug intolerant sustained VT following use of at least one Class III antiarrhythmic as demonstrated by a recurrent arrhythmia and is not a suitable candidate per the investigator's expert opinion for ongoing or alternative drug therapy
4. ECG and/or ICD evidence of a spontaneous VT recurrence within the prior 6 months that is suspected to be the same VT as initially targeted in a prior ablation
5. Subject has minimum 3-month ICD interrogation history available for evaluation
6. Subject has LVEF > 20%, confirmed by echo or comparable technique during baseline evaluation
7. Subject is at least 18 years old
8. Subject has signed the informed consent, and is willing and able to participate in all study procedures and follow up requirements

EXCLUSION CRITERIA:

1. Subjects with VT of idiopathic origin
2. Subjects with VT with ECG or MRI/CT findings suggestive of right ventricular free wall origin
3. Subjects with VTs of septal origin require special care to minimize the risk of heart block, particularly within 2 cm of the AV node/proximal conduction system; Subjects requiring ablation at such locations should only be included when the arrhythmia itself is life-threatening or otherwise sufficiently severe to justify the risk
4. Subject with myocardial infarction (MI) or unstable angina within previous 60 days
5. Subject with cardiac surgery or percutaneous coronary intervention (PCI) within previous 60 days
6. Subject with class IV (NYHA) heart failure
7. Subject with prosthetic cardiac valve(s), severe aortic stenosis or flail mitral valve
8. Subject with left ventricular assist device planned or required for the procedure
9. Subjects with co-morbidities such that they have less than 1-year life expectancy
10. Subject with evidence of intracardiac and/or laminated thrombus (in the left atrium including left atrial appendage or the left ventricle) evident by cardiac CT or transesophageal echo (TEE) and transthoracic echo (TTE) (with contrast if indicated) within 48 hours prior to ablation procedure
11. Subject with thrombocytopenia or other coagulopathy
12. Women who are or may potentially be pregnant (must be post-menopausal or have a negative pregnancy test)
13. Subject with other acute illness or active systemic infection (unrelated to VT or its origin)
14. Significant congenital heart disease or cardiac anomaly
15. Allergy or contraindications to the medications/agents used during a standard ablation/EP intervention.
16. Subject concurrently enrolled in any other investigational drug or device study that the investigator deems would interfere with study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
EFFICACY: Non-inducibility of the targeted clinical VT at end of ablation procedure. | By the end of the procedure
  Completion of intended ablation during treatment setting as measured by non-inducibility of the targeted clinical VT (acute procedural success).
SAFETY: SAEs that are probably or definitely device related within 30 days | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Packer, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Loyola University Medical Center, Maywood, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Vanderbilt Heart, Nashville, Tennessee

REFERENCES:
- [Result] Packer DL, Wilber DJ, Kapa S, Dyrda K, Nault I, Killu AM, Kanagasundram A, Richardson T, Stevenson W, Verma A, Curley M; SERF Investigators. Ablation of Refractory Ventricular Tachycardia Using Intramyocardial Needle Delivered Heated Saline-Enhanced Radiofrequency Energy: A First-in-Man Feasibility Trial. Circ Arrhythm Electrophysiol. 2022 Aug;15(8):e010347. doi: 10.1161/CIRCEP.121.010347. Epub 2022 Jul 1. PMID 35776711